CLINICAL TRIAL: NCT03117530
Title: Targeting Microglial Activation for Treatment of Autism Spectrum Disorder (ASD): A Proof-of-Concept, Target-Engagement Study
Brief Title: Measuring Brain Inflammation in Autism
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: COVID
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Michael Gandal, MD, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-001784
Record Dates: First submitted 2016-11-30; First posted 2017-04-18 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Autism Spectrum Disorder
Keywords: minocycline; brain inflammation; microglia; cognition
MeSH Terms: conditions — Autism Spectrum Disorder; cyclopia sequence; Encephalitis | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Minocycline (Experimental)
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Following initial baseline PET-CT imaging and clinical evaluation, adults with ASD will undergo a 12- week open-label treatment trial of minocycline to be conducted at UCLA under supervision of the UCLA IRB. During weeks 1-6, ASD subjects will be treated with 50 mg minocycline twice daily (low dose). From weeks 7-12, dosing will be increased to 100mg twice daily (typical clinical dosage). Every two weeks during this phase, a treating clinician will measure vital signs, assess safety, record adverse effects, and monitor compliance. Compliance will be obtained as an index of tolerability and will assessed through weekly medication diaries and pill counts.
  Other Names: minocin

SUMMARY:
Autism spectrum disorders (ASD) are highly disabling, persistent neurodevelopmental disorders. There are no available treatments for core symptoms of ASD or biologically-based clinical biomarkers. Emerging evidence indicates that levels of brain inflammation are increased in ASD. In particular, recent work implicates hyperactivity of microglial cells, the resident immune cells of the brain. However, the functional consequences of microglial activation remain unknown. This study will measure microglial activation in ASD using positron emission tomography (PET) brain imaging. Adult males with ASD (n=15) and healthy controls (n=15) will be recruited for this study and undergo comprehensive clinical and behavioral baseline assessment. All subjects will then undergo baseline PET imaging using a radiotracer that labels activated microglia. Subjects with ASD will then undergo 12-week open label treatment with minocycline, an FDA-approved antibiotic thought to block microglial activation. PET imaging will be repeated at 12 weeks to confirm target engagement. A subset of control subjects will also undergo repeat PET imaging to determine test-retest reliability. During minocycline treatment, ASD subjects will be evaluated every 2 weeks for safety, clinical impression, behavioral functioning, and measures of cognition. Results will provide important information regarding the relationship between levels of brain inflammation, cognitive and behavioral function in ASD.

ELIGIBILITY:
Inclusion criteria for participants with ASD

1. Male with a diagnosis of ASD as defined by DSM-5, confirmed by clinical evaluation and ADOS-2.
2. Age 18-35 years inclusive
3. IQ estimate of >70 on VIQ or PIQ
4. Capacity to consent to research
5. Ability to comply with all protocol procedures and assessments
6. Availability of an informant willing to provide information regarding subject behavior and health status (Note: Informant role requires a responsible adult with close, ongoing contact and knowledge of the subject; parent/caregiver acceptable, but not necessary for role)

Exclusion criteria for participants with ASD

1. Evidence of current nicotine, drug, or alcohol abuse or dependence
2. Presence of a chronic medical condition which would potentially influence the assessment of TSPO binding, or interact with study medication (eg. hepatic, neurologic, renal disease) to increase risk to the subject
3. Presence of severe behavioral disturbance likely to require initiation of treatment during the course of the protocol
4. Clinical judgment of the study physician of inability to perform the requirements of the study
5. Current or recent (past 30 days) treatment with minocycline or related compounds, immunosuppressives, or benzodiazepines
6. Homozygous genotype for minor allele of rs6971
7. History of recent febrile illness in past 30 days
8. History of allergic reactions to tetracycline antibiotics
9. Concomitant medication treatment not stable for the 4 weeks prior to study entry or anticipated to change
10. Current prescribed medication likely to confound assessment of TSPO binding

Inclusion criteria for healthy volunteer participants

1. Male in good general health, confirmed by clinical evaluation
2. Age 18-35 years inclusive
3. IQ estimate of >70 on VIQ or PIQ
4. Ability to comply with all protocol procedures and assessments

Exclusion criteria for healthy volunteer participants

1. Diagnosis of an autism spectrum disorder (ASD)
2. Evidence of current nicotine, drug, or alcohol abuse or dependence
3. Presence of a chronic medical condition which would potentially influence the assessment of TSPO binding, or interact with study medication (eg. hepatic, neurologic, renal disease) to increase risk to the subject
4. Presence of current or lifetime severe psychopathology potentially confounding assessment of TSPO binding (psychosis, severe depression, bipolar disorder, Obsessive-Compulsive Disorder)
5. Current prescribed medication likely to confound assessment of TSPO binding
6. Clinical judgment of the study physician of inability to perform the requirements of the study
7. Current or recent (past 30 days) treatment with minocycline or related compounds, immunosuppressives, benzodiazepines, or psychotropic medications likely to confound assessment of TSPO binding
8. Homozygous genotype for minor allele of rs6971
9. SRS-2 T-score score of >59
10. History of recent febrile illness in past 30 days

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-04-11 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate differences in CNS microglial activation in adults with ASD versus healthy volunteers via in vivo CNS binding of [11C]-DAA1106 | Data will be collected at PET scan #1, which will take place during screening (Days -28 to 0) for the study
Evaluate the effect of 12-weeks of minocycline exposure on CNS microglial activation in adults with ASD by measuring change in [11C]-DAA1106 binding pre- and post- treatment | Data will be collected at PET scan #1 (between days -28 and 0 before intervention) and at PET scan #2 during Week 12 of intervention

SECONDARY OUTCOMES:
Effect of minocycline exposure on cognition across seven cognitive domains before and after low dose intervention and regular dose intervention as measured by MCCB (MATRICS Consensus Cognitive Battery) subdomain scores | Data will be collected at baseline and during Weeks 6 and 12 of intervention
Effect of minocycline exposure on self-rated anxiety and emotion regulation as measured by ADAMS (Anxiety and Depression Mood Scale) | Data will be collected at baseline and during Weeks 6 and 12 of intervention
Effect of minocycline exposure on peripheral inflammatory cytokine profiles as measured by DNA and RNA expression in blood samples | Data will be collected PET #1 (week 0) and at PET scan #2 (Week 12)

OTHER OUTCOMES:
Change in clinician-rated global improvement as measured by CGI | Data will be collected at Screening Visit #1 (between days -28 and 0 before intervention) and at visits during Weeks 6 and 12 of intervention
Change in self-reported symptoms of ASD with minocycline treatment as measured by SRS-2 | Data will be collected at Screening Visit #1 (between days -28 and 0 before intervention) and at visits during Weeks 6 and 12 of intervention
Change in informant-reported symptoms of ASD with minocycline treatment as measured by ABC-CV | Data will be collected at Screening Visit #1 (between days -28 and 0 before intervention) and at visits during Weeks 6 and 12 of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gandal, MD PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared